CLINICAL TRIAL: NCT06503809
Title: Efficacy and Safety of a Ketogenic Diet in Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202305041
Record Dates: First submitted 2024-06-27; First posted 2024-07-16 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; Ketogenic diet; Insulin sensitivity; Continuous glucose monitoring; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Hypoglycemia | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic Diet (Experimental): The Ketogenic Diet group will consume a very-low carbohydrate diet (<50 g/day) diet. Participants will receive isocaloric packed-out meals for 12 weeks.
  Interventions: Behavioral: Ketogenic Diet
- Standard Care (Active Comparator): The Standard Care group will consume a diet consistent with the guidelines recommended by the American Diabetes Association that is high in non-starchy vegetables and lean protein sources and low in added sugar. Participants will receive isocaloric packed-out meals for 12 weeks.
  Interventions: Behavioral: Standard Diet

INTERVENTIONS:
Behavioral: Ketogenic Diet — Participants will consume a very-low-carbohydrate ketogenic diet for 12 weeks.
  Arms: Ketogenic Diet
Behavioral: Standard Diet — Participants will consume an American Diabetes Association-recommended standard diet for 12 weeks.
  Arms: Standard Care

SUMMARY:
Despite strong evidence that tight control of blood sugar reduces the risk of diabetes complications, most people with type 1 diabetes do not achieve recommended blood sugar targets. This randomized controlled trial will test whether a very-low- carbohydrate ketogenic diet can effectively and safely improve blood sugar control in adults with type 1 diabetes.

DETAILED DESCRIPTION:
A very-low-carbohydrate ketogenic diet (≤50 g carbohydrate/day) could reduce glycemic variability, total daily insulin requirement, and HbA1c in people with type 1 diabetes (T1D). Indeed, several case series and observational studies of using a ketogenic diet (KD) in people with T1D have observed such benefits. However, no randomized controlled trials (RCTs) have evaluated the efficacy of KD for >7 days in people with T1D. In addition, there are serious concerns regarding the safety and tolerability of a KD in patients with T1D, including the potential for an increased risk of hypoglycemia, diabetic ketoacidosis, dyslipidemia, insulin resistance, decreased bone mineral density, and impaired quality of life. This study is a 12-week RCT to evaluate the clinical efficacy, metabolic function, safety, socio-behavioral impact, acceptability and potential for dissemination of an isocaloric KD compared with an American Diabetes Association-recommended control diet in adults with T1D.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤65 years
* T1D diagnosed >1 year prior to screening
* HbA1c 7.0%-9.0%
* Stable insulin delivery method for the past 30 days
* Ability to read all device instructions and insulin pump settings
* eGFR ≥60 mL/min/1.73 m2
* Use of an insulin pump or insulin delivery by multiple daily injections
* Use of personal CGM for at least 12 weeks and willing to change to Dexcom CGM for the duration of the study, if using a different sensor, to reduce variability in glucose values associated with different CGM products
* Use of cellular phone with data capability for wireless connectivity to the CGM system.

Exclusion Criteria:

* Body mass index <20.0 or >34.9 kg/m2
* Severe gastroparesis or history of bariatric surgery
* Diabetes-related hospitalization (including for diabetic ketoacidosis or severe hypoglycemia) within 12 months of screening
* Poorly controlled hypertension (SBP ≥160 mmHg or DBP ≥100 mmHg)
* Taking diabetes medications, other than insulin (particularly SGLT2 inhibitors, which are associated with an increased risk of euglycemic DKA)
* Structured exercise >210 minutes per week
* Pregnant, lactating, not using effective birth control if premenopausal, or planning to become pregnant within the 6-month study period
* Unstable weight (>4% change in the last 2 months)
* Significant organ system dysfunction (e.g., severe pulmonary, renal, hepatic, or cardiovascular disease)
* Anemia (Hgb <10 g/dL)
* Major psychiatric illness
* Active tobacco use (>8 cigarettes/day) or illegal drug use
* Regular alcohol consumption (>10 standard drinks per week)
* Use of medications known to affect the study outcome measures or increase the risk of study procedures that cannot be temporarily discontinued for this study
* Familial hypercholesterolemia
* Active eating disorder
* Dietary restrictions incompatible with a very-low-carbohydrate KD, vegan diet, vegetarian diet, severe lactose intolerance, severe aversion/sensitivity to eggs, fish, nuts, wheat, or soy, and any anaphylactic food allergy
* Already consuming a low-carbohydrate (<130 g/day) diet
* Persons who are not able to grant voluntary informed consent
* Persons who are unable or unwilling to follow the study protocol or who, for any reason, the research team considers an inappropriate candidate for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in continuous glucose monitor (CGM) time-in-range | Before and immediately after the dietary intervention
  Interstitial glucose percent time in range assessed by using a continuous glucose monitor
Change in skeletal muscle insulin sensitivity | Before and immediately after the dietary intervention
  Insulin sensitivity will be determined by the hyperinsulinemic-euglycemic clamp procedure

SECONDARY OUTCOMES:
Change in daily insulin requirements | Assessed before, during, and immediately after the dietary intervention
  The daily total dose of insulin used will be assessed
Change in 24-hour glucose concentrations | Before and immediately after the dietary intervention
  Plasma glucose concentrations will be evaluated from frequent blood samples over a 24 hour period
Change in 24-hour glucagon concentrations | Before and immediately after the dietary intervention
  Plasma glucagon concentrations will be evaluated from frequent blood samples over a 24 hour period
Change in whole-body palmitate turnover | Before and immediately after the dietary intervention
  Palmitate turnover will be measured by isotope dilution
Change in plasma lipid profile | Before and immediately after the dietary intervention
  Fasting plasma lipid profile will be assessed
Change in hepatic de novo lipogenesis | Before and immediately after the dietary intervention
  Hepatic de novo lipogenesis will be assessed by the deuterated water method
Change in de novo cholesterol synthesis | Before and immediately after the dietary intervention
  Cholesterol synthesis will be assessed by the deuterated water method
Change in fat mass | Before and immediately after the dietary intervention
  Fat mass will be assessed using dual-energy x-ray absorptiometry (DXA)
Change in fat-free mass | Before and immediately after the dietary intervention
  Fat-free mass will be assessed using dual-energy x-ray absorptiometry (DXA)
Change in intrahepatic triglyceride content | Before and immediately after the dietary intervention
  Intrahepatic triglyceride content will be assessed by magnetic resonance imaging (MRI)
Change in specific adipose tissue volumes | Before and immediately after the dietary intervention
  Specific adipose tissue depot volumes will be assessed by magnetic resonance imaging (MRI)
Change in plasma hs-CRP | Before and immediately after the dietary intervention
  Plasma hs-CRP will be measured
Change in plasma PAI-1 | Before and immediately after the dietary intervention
  Plasma PAI-1 will be measured
Change in plasma IL-6 | Before and immediately after the dietary intervention
  Plasma IL-6 will be measured
Change in plasma TNF-alpha | Before and immediately after the dietary intervention
  Plasma TNF-alpha will be measured
Change in plasma markers of liver function | Before and immediately after the dietary intervention
  Plasma markers of liver function will be measured
Change in plasma markers of kidney function | Before and immediately after the dietary intervention
  Plasma markers of kidney function will be measured
Change in plasma markers of bone turnover | Before and immediately after the dietary intervention
  Plasma markers of bone turnover will be measured
Change in percent time in hypoglycemia | Before and immediately after the dietary intervention
  Percent time in hypoglycemia will be assessed by using a continuous glucose monitor
Change in percent time in hyperglycemia | Before and immediately after the dietary intervention
  Percent time in hyperglycemia will be assessed by using a continuous glucose monitor
Level 3 hypoglycemia event rate | During the dietary intervention
  Number of event rates for level 3 hypoglycemia defined as blood glucose or sensor glucose concentration <54 mg/dL with neurological symptoms of low blood glucose concentration such as confusion, lethargy, seizure, or coma
Diabetic ketoacidosis event rate | During the dietary intervention
  Number of diabetic ketoacidosis event rates defined as plasma beta-hydroxybutyrate concentration >3 mmol/L, plasma bicarbonate concentration < 18 mmol/L, pH<7.30, and symptoms including polyuria, polydipsia, nausea, vomiting, or abdominal pain
Change in bone mineral density | Before and immediately after the dietary intervention
  Bone mineral density will be assessed using dual-energy x-ray absorptiometry (DXA)
Change in sociobehavioral factors | Before and immediately after the dietary intervention
  Sociobehavioral factors will be assessed by using validated questionnaires
Knowledge and perceptions of the diet | Immediately after the dietary intervention
  Dissemination and implementation (D&I) survey measures available from the Washington University Center for Diabetes Translation Research D&I Core will be used to assess participants' knowledge and perceptions of the diets at the end of the study
Adaptations needed to implement the diet at the population level | Immediately after the dietary intervention
  Qualitative interviews will be performed to understand perceptions of the diet interventions and what adaptations might be needed to disseminate the intervention at a population level
Change in glycated hemoglobin and albumin | Before, during, and immediately after the dietary intervention
  Glycated hemoglobin and albumin will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States